CLINICAL TRIAL: NCT05737160
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Phase III Study of Telitacicept in Patients With Generalized Myasthenia Gravis
Brief Title: Study of Telitacicept in Generalized Myasthenia Gravis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18C029
Record Dates: First submitted 2023-02-12; First posted 2023-02-21 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2024-10

CONDITIONS: Myasthenia Gravis, Generalized
Keywords: Myasthenia Gravis; Autoimmune Diseases; Muscle Weakness
MeSH Terms: conditions — Myasthenia Gravis; Autoimmune Diseases; Muscle Weakness | interventions — telitacicept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telitacicept (Experimental): Participants will receive subcutaneous Telitacicept 240 mg once a week for a total of 48 doses in addition to MG SoC.
  Interventions: Biological: Telitacicept
- Placebo (Placebo Comparator): Participants will receive subcutaneous placebo once a week for a total of 24 doses (part A) and then weekly subcutaneous Telitacicept 240 mg for 24 doses (part B) in addition to MG SoC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Telitacicept — Administered as an SC infusion
  Other Names: RC18
  Arms: Telitacicept
Drug: Placebo — Administered as an SC infusion
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Telitacicept in the treatment of patients with generalized myasthenia gravis.

DETAILED DESCRIPTION:
This study consists of a screening period, a double-blind treatment period (part A) and an open-label treatment period (part B). After screening, eligible subjects will be randomized in a 1: 1 ratio to receive either subcutaneous Telitacicept 240 mg or placebo once a week for 24 doses (part A). Completing part A, subjects will automatically enter part B. In part B, all subjects will receive weekly subcutaneous Telitacicept 240 mg for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent provided;
2. Male or female patients aged 18-80 years;
3. Diagnosis with generalized myasthenia gravis;
4. MGFA Class II, III, or IVa;
5. AChR-Ab or MuSK-Ab positive;
6. A total MG-ADL score of ≥ 6 with less than 50% of the total score due to ocular symptoms;
7. QMG ≥ 8, with ≥ 4 items score at least 2;
8. Have been on a stable MG SoC regimen.

Exclusion Criteria:

1. Patients with autoimmune diseases other than MG;
2. Abnormal laboratory results；
3. Use of immunosuppressants other than standard therapy within 1 month before randomization;
4. Use of biologic agents targeting therapy, such as Rituximab or complement C5 inhibitors, within 6 months before randomization;
5. Use of neonatal Fc receptor (FcRn) antagonists, intravenous immunoglobulin (IVIg), or plasmapheresis within 2 months before randomization;
6. Significant cardiovascular disease, liver, kidney, respiratory, endocrine or hematologic disease, or other medical conditions that, in the opinion of the investigator, would preclude the subject's participation in the study or require hospitalization during the study;
7. Acute or chronic infection requiring treatment;
8. Current active hepatitis;
9. HIV antibody positive;
10. Patients currently suffering from thymoma-associated immunodeficiency syndrome (Good's syndrome) or who underwent thymectomy within 6 months before screening;
11. Received or plan to receive any live vaccine within 3 months prior to randomization;
12. Patients with malignant tumors;
13. Allergy to biological products of human origin;
14. Participation in any clinical trial 28 days prior to randomization or within 5 times the half-life of an investigational drug (whichever is longer);
15. Pregnant or lactating women, and those intending to become pregnant during the trial;
16. Patients considered unsuitable by the investigator to participate in the trial (e.g., patients with severe mental disorders);

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in MG-ADL | Week 24
  The MG-ADL is an 8-item patient-reported scale that measures MG symptoms and functional status. Each item ranges from 0 to 3 for a total score range of 0 to 24.

SECONDARY OUTCOMES:
Change from baseline in MG-ADL | Weeks12, 36, 48
  The MG-ADL is an 8-item patient-reported scale that measures MG symptoms and functional status. Each item ranges from 0 to 3 for a total score range of 0 to 24.
Change from baseline in QMG | Weeks 12, 24, 36, 48
  The quantitative myasthenia gravis (QMG) score is a 13-item scale used to quantify disease severity in myasthenia gravis (MG). Total QMG score ranges from 0 (no myasthenic findings) to 39 (maximal myasthenic deficits).
Proportion of subjects with ≥ 3 points reduction from baseline in MG-ADL | Weeks 24, 48
  The MG-ADL is an 8-item patient-reported scale that measures MG symptoms and functional status. Each item ranges from 0 to 3 for a total score range of 0 to 24.
Proportion of subjects with a decrease of ≥ 5 points from baseline in QMG | Weeks 24, 48
  The quantitative myasthenia gravis (QMG) score is a 13-item scale used to quantify disease severity in myasthenia gravis (MG). Total QMG score ranges from 0 (no myasthenic findings) to 39 (maximal myasthenic deficits).

CONTACTS AND LOCATIONS:
Locations (51):
- China (51):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - Beijing Hospital, Beijing, Beijing Municipality
  - Xuanwu Hospital of Capital Medical University, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Nanyang First People's Hospital, Nanyang, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Wuhan Hospital of Traditional Chinese and Western Medicine (Wuhan No.1 Hospital), Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Inner Mongolia Autonomous Region People's Hospital, Hohhot, Inner Mongolia
  - Nanjing First Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - Dalian Municipal Central Hospital, Dalian, Liaoning
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - The Second Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - The First Affiliated Hospital of Jinzhou Medical University, Jinzhou, Liaoning
  - Shengjing Hospital Affiliated to China Medical University, Shenyang, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The People's Hospital of Liaoning Province, Shenyang, Liaoning
  - The Second Affiliated Hospital of PLA Air Force Military Medical University, Xi'an, Shaanxi
  - Xi'an Hi-tech Hospital, Xi'an, Shaanxi
  - Xianyang Hospital of Yan'an University, Xianyang, Shaanxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Jining No.1 People's Hospital, Jining, Shandong
  - Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi
  - The First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Affiliated Hospital of North Sichuan Medical College, Nanchong, Sichuan
  - First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The First People's Hospital of Yunnan Province, Kunming, Yunnan
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Sir Run Run Shaw Hospital, affiliated with to Zhejiang University College of Medicine, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang